CLINICAL TRIAL: NCT02569294
Title: Feasibility and Impact of Yoga, Self-hypnosis and Cognitive-behavioral Group Interventions in Improving Well-being of Breast Cancer Patients
Brief Title: Feasibility and Impact of Group Interventions on Breast Cancer Patients Well-being
Acronym: GIBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Isabelle Bragard, Ph.D., University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Y-HYP-CBT-037
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: group interventions; emotional distress; breast cancer; yoga; hypnosis; cognitive-behavioral therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Choice 1: Yoga intervention (Experimental): See intervention description
  Interventions: Behavioral: Yoga intervention
- Choice 2: Hypnosis intervention (Experimental): See intervention description
  Interventions: Behavioral: Hypnosis intervention
- Choice 3: CBT intervention (Experimental): See intervention description
  Interventions: Behavioral: CBT intervention
- Control group (No Intervention): Participants who agreed not to participate in any of the interventions proposed.

INTERVENTIONS:
Behavioral: Yoga intervention — Hatha-yoga intervention included 6 weekly 90-min sessions in groups of 3 to 8 participants led by Hatha-yoga trained teachers. This program was developed previously in Montreal and the following were included at each session: 1) preparatory warm-up synchronized with breathing; 2) selected postures (e.g. forward , backward-, and side-bending asanas in sitting and lying positions); 3) deep relaxation; 4) alternate-nostril breathing or pranayama; and 5) meditation. Each participant received a DVD to encourage at-home practice.
  Arms: Choice 1: Yoga intervention
Behavioral: Hypnosis intervention — Hypnosis intervention included 6 sessions of 2 hours every 2 weeks. This was led by an anesthesist with experience in oncology and trained in hypnosis. Based on years of consultation with cancer patients, her team created a negotiating approach that fosters shared decision-making through using tasks that are centered on general well-being rather than on the health problem itself. Patients were asked to be actively involved. Several topics are addressed through tasks: eg. adjusting self-expectations. Patients were also required to keep a work-diary that was reviewed at the beginning of each session. At the end of the session, a 15-min hypnosis exercise is conducted. They receive CDs containing the hypnosis exercises and homework assignments.
  Arms: Choice 2: Hypnosis intervention
Behavioral: CBT intervention — CBT intervention included 6 weekly 90-min sessions in groups of 3 to 8 participants led by CBT-trained psychologists with experience in psycho-oncology. This program was developed by team leaders and is modelled on the work of Andersen et al. (2008) and Savard (2010). The intervention targets were: 1) breast cancer, meaning of illness, understanding stress and responses to it; 2) impact of treatment on body image; 3) impact of treatment on self-esteem; 4) fear of recurrence; 5) relationships with relatives and health professionals; and 6) life projects, return to daily activities and work. Relaxation training took place at the end of each session and participants performed tasks between sessions.
  Arms: Choice 3: CBT intervention

SUMMARY:
This is a clinical non-randomized prospective study. This study had two objectives. The fist one was to determine the interest of breast cancer patients in participating in one of three group interventions (CBT, yoga or self-hypnosis) by assessing the participation rate, the reasons for choosing a particular group or decline the offer. The second objective was to evaluate and compare the benefits of these three interventions on emotional distress, QoL, sleep quality and mental adjustment to cancer, at three times after the end of the interventions (just after the end, at a 3-month and at a 9-month follow-up).

DETAILED DESCRIPTION:
This study had two objectives. The fist one was to determine the interest of breast cancer patients in participating in one of three group interventions (cognitive-behavioral therapy, yoga or self-hypnosis) by assessing the participation rate, the reasons for choosing a particular group or decline the offer. The second objective was to evaluate and compare the benefits of these three interventions on emotional distress, QoL, sleep quality and mental adjustment to cancer.

Eligible breast cancer patients were identified through an institutional database or by referring physicians and were approached by phone to inform them of the intervention. They were given a choice between the three group interventions: CBT, yoga and self-hypnosis. Patients who agreed not to participate in any of the interventions were included in the control group. After giving written informed consent, patients completed a baseline assessment including self-reported measures. Follow-up assessment was conducted one week after the group intervention, and at a 3-month and 9-month follow-up. Interventions were proposed according to previous results showing the patient's interest in CBT, yoga and self-hypnosis, and the expertise of the team. Each intervention included 6 sessions of 1.5 hours.

The primary outcome measure was the interest in the three interventions (participation rate in each group). Since the study was first designed to determine interest, no sample size calculation was performed. Secondary outcomes were responses concerning emotional distress, QoL, sleep quality and mental adjustment to cancer assessed with self-reported questionnaires before and after the group interventions.

Descriptive statistics (percentages, means and standard deviation (SD)) were used to describe the proportions of patients who were interested in the group interventions and to examine their demographic, medical and psychological data. Baseline time 0 demographic, medical and psychological data were compared between groups to test for initial group equivalency using inferential statistics: analysis of variance (ANOVA) and Chi-square test, as appropriate. To be considered for the data analysis, patients had to attend at least three sessions. Multivariate analyses were calculated regarding group interventions and time of medical treatments (during or after chemo/radiation therapy). The pre- and post-assessment comparison of each measure within each group was made using the Wilcoxon test for matched pairs. All statistical tests were two-tailed, and a P-value <0.05 was considered statistically significant. Investigators also calculated Cohen's d effect size for each group. The analyses were performed with SPSS Version 21.0 (IBM Corp., Armonk, N.Y).

ELIGIBILITY:
Inclusion Criteria:

* first breast cancer without metastases
* between 18 and 75-year-old
* ability to read, write and speak French.

Exclusion Criteria:

* Patients with a diagnosed psychiatric disorder or dementia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Interest of patients in the three groups | 3 years
  The first outcome is to determine the interest of breast cancer patients in participating in one of three group interventions (CBT, yoga or self-hypnosis) by assessing the participation rate in each group (N and %).
Reasons for choosing a particular group | 3 years
  The second outcome is to determine the reasons for choosing a particular group (open question).
Reasons for declining to participate | 3 years
  The third outcome is to determine the reasons for declining to participate to the groups (open question).

SECONDARY OUTCOMES:
Emotional distress | 4 years
  This outcome is measured with the Hospital Anxiety Depression Scale (HADS) at 4 time periods: before and just after the intervention, at a 3-month and a 9-month follow-up. The HADS is a reliable and validated 14-item measure assessing anxiety and depression in physically ill subjects [27]. Seven items for anxiety and 7 for depression are rated on a 4-point Likert scale (0=symptom not present to 3=symptom considerable). Each subscale is scored from 0 to 21 (0-7: 'normal range', 8-10: 'borderline', 11-21: 'probable presence of anxiety or depressive disorder').
Quality of Life | 4 years
  This outcome is measured with European Organization for Research and Treatment of Cancer-Quality of Life Core Questionnaire-30 (EORTC-QLCQ30) and the Breast-cancer specific module (BR23) at 4 time periods: before and just after the intervention, at a 3-month and a 9-month follow-up.
Mental adjustment to cancer | 4 years
  This outcome is measured with the Mental Adjustment to Cancer Scale (MAC) at 4 time periods: before and just after the intervention, at a 3-month and a 9-month follow-up. This is a 40-item questionnaire addressing reactions of patients on having cancer. Items are given as statements, and patients assess their agreement using a 4-point Likert-scale ('definitely does not apply to me' to 'definitely applies to me'). There are five subscales: Fighting Spirit (cut-off ≥47); Helplessness/Hopelessness (cut-off ≥11); Anxious Preoccupation (cut-off ≥25); Fatalism (cut-off ≥22) and Avoidance (cut-off ≥3); and two general subscales: Summary Positive Adjustment Scale (cut-off ≥47) and Summary Negative Adjustment Scale (cut-off ≥36).
Quality of sleep | 4 years
  This outcome is measured with the Insomnia Severity Index (ISI) at 4 time periods: before and just after the intervention, at a 3-month and a 9-month follow-up. This is a 7-item measure of subjective sleep complaints and associated distress. Items are scored on a 5-point Likert scale ranging from 0 to 4 with higher scores representing more severe insomnia symptoms. The cut-off scores are 0-7 (no clinically significant sleep difficulties), 7-14 (sleep difficulties warrant further investigation) and 15+ (presence of clinically significant insomnia).

CONTACTS AND LOCATIONS:
Overall Officials: Guy Jerusalem, Prof., Study Director — University of Liege
Locations (1):
- University Hospital of Liege, Liège, Belgium

REFERENCES:
- [Derived] Gregoire C, Nicolas H, Bragard I, Delevallez F, Merckaert I, Razavi D, Waltregny D, Faymonville ME, Vanhaudenhuyse A. Efficacy of a hypnosis-based intervention to improve well-being during cancer: a comparison between prostate and breast cancer patients. BMC Cancer. 2018 Jun 22;18(1):677. doi: 10.1186/s12885-018-4607-z. PMID 29929493